CLINICAL TRIAL: NCT01261299
Title: A Phase 0 Clinical Trial of Microdosing Carboplatin and Molecular Profiling for Chemoresistance
Brief Title: Clinical Study of Microdosing Carboplatin in Lung or Bladder Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Contract ended
Sponsor: University of California, Davis (Other)
Collaborators: Lawrence Livermore National Laboratory (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#200; 201018146 (Other: UC Davis)
Record Dates: First submitted 2010-12-09; First posted 2010-12-16 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms
Keywords: Phase 0 Clinical trial; Human microdosing trial; Drug resistance, neoplasm; Carcinoma, Non-small cell lung; Urinary Bladder Neoplasm; Individualized Medicine; Carboplatin; Carboplatin-DNA adducts
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carbon-14-labeled carboplatin (Experimental): Patients are eligible for this study if they have non-small cell lung cancer or bladder cancer and will receive cisplatin or carboplatin-based chemotherapy for the treatment of cancer. They will receive one microdose of C-14-carboplatin approximately 4 hours before scheduled biopsy/surgery. One blood draw and a few milligrams of leftover tumor tissue will be taken for analysis of carboplatin-DNA adduct levels. The dose of carboplatin will be about 1/100th the therapeutic dose.
  Interventions: Drug: Carbon-14-labeled carboplatin

INTERVENTIONS:
Drug: Carbon-14-labeled carboplatin — Patients are eligible for this study if they have non-small cell lung cancer or bladder cancer and will receive cisplatin or carboplatin-based chemotherapy for the treatment of cancer. They will receive one microdose of C-14-carboplatin approximately 4 hours before scheduled biopsy/surgery. One blood draw and a few milligrams of leftover tumor tissue will be taken for analysis of carboplatin-DNA adduct levels. The dose of carboplatin will be about 1/100th the therapeutic dose.

SUMMARY:
Carboplatin kills cancer cells mainly through induction of DNA damage (drug-DNA adducts). The goal of this clinical trial is to determine if chemoresistance to carboplatin can be identified by measuring carboplatin-induced DNA monoadducts, the precursor of Pt-DNA diadducts or crosslinks, from subtherapeutic drug doses given prior to the initiation of chemotherapy. We hypothesize that low levels of carboplatin-DNA monoadducts and rapid drug-DNA adduct repair correlate with chemoresistance. A highly sensitive technology, called accelerator mass spectrometry (AMS), will be used to measure carboplatin-DNA monoadducts from patient samples. AMS can measure C-14 at the attomole level in specimens of milligram size. In this study, patients will receive one non-toxic "microdose" (defined as 1/100th the therapeutic dose) of C-14-labeled carboplatin. Blood specimens will be drawn for determination of carboplatin-DNA monoadduct formation and repair in peripheral blood mononuclear cells (PBMC), and pharmacokinetics (PK) will be determined from serum ultrafiltrate. In patients microdosed prior to providing tumor samples, a few milligrams of leftover tumor biopsy/resection specimens will be analyzed for formation of carboplatin-DNA monoadducts. Patients will subsequently receive carboplatin-based chemotherapy. The levels of microdose-induced carboplatin-DNA monoadducts will be correlated with response to chemotherapy. Some blood and biopsy samples will be assayed by RT-PCR for several putative resistance markers at the mRNA level. Side effects will also be monitored and compared to the AMS data. This trial will also utilize PK, DNA repair and pharmacogenomics data in order to determine some of the underlying chemoresistance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have clinical diagnosis of lung or bladder cancer. The term "clinical diagnosis" means that patients are diagnosed with NSCLC or bladder transitional cell carcinoma (TCC) based on imaging studies, but will need further biopsy/resection to obtain tissue in order to confirm the diagnosis. However, some patients may not have cancer as determined by pathology examination of the tissue, or may have a different cancer after biopsy/resection is performed. If the diagnosis of NSCLC or bladder cancer is confirmed, platinum-based chemotherapy must be planned either for neoadjuvant chemotherapy for Stage II or above bladder cancer, or palliative therapy for stage III or IV lung or bladder cancer regardless of patient participation in this study. Stage II or above TCC patients and stage IV NSCLC patients that will receive platinum-based chemotherapy will be eligible for this study. Patients with Stage III or IV lung or bladder cancer must have measurable lesion(s).
* Prior radiation or surgery is allowed, but should be finished at least 2 weeks prior to study enrollment. If a participant has prior radiation therapy, at least one measurable lesion outside of the radiation field should be available for the evaluation of response to chemotherapy.
* Participants must be 18 years or older. We do not see any patients with NSCLC or bladder TCC are diagnosed under the age of 18 years.
* ECOG performance status equal or less than to 2 (Karnofsky equal to or greater than 50%).
* Life expectancy of at least 3 months.
* Participants must have normal organ and marrow function as defined below: Absolute neutrophil count greater than/equal to 1,500/microL; Platelet count greater than/equal to 100,000/microL; Total bilirubin less than 1.5 X ULN; AST (SGOT) less than/equal to 2.5 X ULN; Creatinine less than 1.5 X ULN
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after study participation.
* Ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients must not receive concomitant radiation with chemotherapy if they do not have any measurable lesions outside of the radiation field.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants who are pregnant or nursing.
* Participants who are allergic to platinum agents.
* Participants who receive chemotherapy before that includes cisplatin, carboplatin or oxaliplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Correlation of carboplatin-DNA monoadducts induced by microdoses of carboplatin with cancer response to carboplatin-based chemotherapy | Patients will be evaluated for response to chemotherapy after they have received 2 to 3 cycles of chemo that is about 6-9 weeks after treatment is started.
  Imaging studies (including CT, MRI, PET/CT and CXR) and cystoscopy will be performed to evaluate the response. The RECIST 1.1 will be used to determine the cancer response. Tumor response, including complete response (CR, or complete disappearance) or partial response (PR, at least a 30% decrease of target lesion) will be correlated with the patient's carboplatin-DNA monoadduct levels.

SECONDARY OUTCOMES:
Determination of the underlying chemoresistance mechanisms to carboplatin | The chemoresistance mechanisms will be determined from the time of this microdosing study to the time patients receive 2 to 3 cycles of chemo that is about 6-9 weeks after treatment is started.
  The half-life of carboplatin and the repair rate of DNA monoadducts (decrease of DNA monoadducts over 24 hours) in PBMC and tumor tissue will be determined and calculated. The ERCC1 expression levels will be determined with quantitative RT-PCR using beta-actin as the internal control. These parameters will be correlated with tumor response (CR or PR) to chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chong-xian Pan, MD, PhD, Study Chair — University of California, Davis
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California